CLINICAL TRIAL: NCT04827693
Title: The Cortical Shield for Facial Bone Reconstruction of Severely Damaged Sockets With Simultaneous Implant Placement
Brief Title: The Cortical Shield for Facial Bone Reconstruction
Status: Completed | Type: Observational
Sponsor: Verdugo, Fernando, DDS (Individual)
Responsible Party: Sponsor
Other Study IDs: Ver152007
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Tooth Loss; Tooth Diseases; Tooth Fracture; Tooth Injuries; Periodontal Bone Loss; Periodontitis; Peri-Implantitis; Tooth Decay
Keywords: tooth socket; bone grafting; bone regeneration; dental implant; osseointegration
MeSH Terms: conditions — Tooth Loss; Tooth Diseases; Tooth Fractures; Tooth Injuries; Alveolar Bone Loss; Periodontitis; Peri-Implantitis; Dental Caries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Immediate: implants are placed immediately after tooth extraction
- Delayed: implants are placed months after the tooth has been extracted

SUMMARY:
To evaluate a novel technique of bone regeneration and simultaneous implant placement in severely damaged sockets.

DETAILED DESCRIPTION:
Patients requiring a single implant, presenting severe facial bone loss as a result of previous infection, failed socket grafting or trauma, will enter this cross-sectional study. Socket reconstruction and simultaneous implant placement will be performed through periosteal-guided bone regeneration (PGBR). Implant timing: immediate or delayed. Implants will be encased in a customized shield of autogenous cortical bone harvested from an adjacent site. A re-entry surgery will be performed at 12-17-weeks to evaluate bone regeneration. Peri-implant tissues will be assessed following established success criteria. Implants will be evaluated for the presence of Periimplantitis.

ELIGIBILITY:
Inclusion Criteria:

* ASA1 or ASA2 (American Society of Anesthesiologists)
* Healthy individuals with good oral hygiene and motivation
* No systemic uncontrolled diseases
* Not taking drugs known to modify bone metabolism

Exclusion Criteria:

* Individuals with untreated & generalized severe periodontitis
* Heavy smokers (>10 cigarettes/day)
* Poor oral hygiene
* Diabetes (HbA1C >6.5% as cutoff value)
* Uncontrolled cardiovascular disease
* Poor overall health (ASA IV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients requiring single implants to replace missing teeth to restore masticatory function and esthetics. Options of immediate or delay placement will be chosen based on the current status of the site to be restored at the time of referral.
  The present cross-sectional quasi-experimental study is conducted in a specialty clinic in accordance to the requirements of the 1964 Helsinki Declaration
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-04-05 (Actual)

PRIMARY OUTCOMES:
Individuals presenting alveolar Facial Bone regeneration at re-entry | 1 year
  Bone regeneration of the dent-alveolar socket

SECONDARY OUTCOMES:
Pink Esthetic Scores | 1 year
  Scores 1-10: the higher the score the better the esthetic outcome. Evaluates soft tissue esthetics around the regenerated bone & implant: mesial & distal papillae, curvature of facial mucosa, level of facial mucosa, root convexity/soft tissue color & texture
Facial implant transparency | 1 year
  Presence of implant transparency at 1 year follow-up: Yes/No
Band of Keratinized tissue | 1 year
  Evaluation of the presence of a band of keratinized tissue around the implant: > 2mm or < 2mm
Implant crestal bone loss | 1 year
  Radiographic evaluation of peri-implant marginal crestal bone loss

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Verdugo, PhD, Principal Investigator — University of Sacro Cuore
Locations (1):
- Fernando Verdugo, DDS, Corp, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No